CLINICAL TRIAL: NCT06775093
Title: Effects of GLP-1 Receptor Agonists Combined with Metformin and Healthy Lifestyle Education Prior to Fertility Treatment on Reproductive Outcomes in Women with PCOS and Obesity
Brief Title: Effects of GLP-1RAs on Reproductive Outcomes in PCOS and Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jie Qiao, Dean, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2024472
Record Dates: First submitted 2025-01-04; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Polycystic Ovary Syndrome; Obesity; Infertility, Female
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Infertility, Female | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 RAs combined with metformin and healthy lifestyle education (Experimental): Benaglutide injection (Fisuomei®, National Medicine Standard No. S20230042, Shanghai Renhui Biopharmaceutical Co., Ltd.) was administered at an initial dose of 0.06 mg per injection, three times daily, via subcutaneous injection 5 minutes before meals. After establishing tolerance, the dose was increased weekly by 0.04 mg per injection, reaching 0.2 mg per injection after four weeks, administered three times daily for a total of 12 weeks. Metformin hydrochloride (Glucophage®, National Medicine Standard No. H20023370, Shanghai Bristol-Myers Squibb Pharmaceuticals Co., Ltd.) was prescribed at a dose of 0.5 g twice daily for 12 weeks, taken with meals. After 12 weeks of treatment or achieving a 10% reduction in baseline body weight, the medications were discontinued. Patients were advised to maintain a healthy diet and engage in appropriate physical activity. Assisted pregnancy treatments were initiated 4 weeks after completing the weight loss phase.
  Interventions: Drug: GLP-1 receptor agonist; Drug: Metformin; Behavioral: healthy lifestyle education
- metformin and healthy lifestyle education (Active Comparator): Metformin hydrochloride (Glucophage®, National Medicine Standard No. H20023370, Shanghai Bristol-Myers Squibb Pharmaceuticals Co., Ltd.) was administered at a dose of 0.5 g twice daily for 12 weeks, taken with meals. After 12 weeks of treatment or achieving a 10% reduction in baseline body weight, the medication was discontinued. Patients were instructed to maintain a healthy diet and engage in appropriate physical activity. Assisted pregnancy treatment was initiated 4 weeks after completing the weight loss phase.
  Interventions: Drug: Metformin; Behavioral: healthy lifestyle education

INTERVENTIONS:
Drug: GLP-1 receptor agonist — 3 months
  Other Names: Benaglutide
  Arms: GLP-1 RAs combined with metformin and healthy lifestyle education
Drug: Metformin — 3 months
Behavioral: healthy lifestyle education — 3 months

SUMMARY:
The goal of this clinical trial is to examine whether benalutide combined with metformin and healthy lifestyle education in women with PCOS and obesity prior to fertility treatment improves live birth rate and other reproductive, maternal and perinatal outcomes compared to metformin plus healthy lifestyle education.

DETAILED DESCRIPTION:
Benalutide, a short-acting recombinant human GLP-1RAs with nearly 100% homology to human GLP-1, has been approved by the Chinese National Medical Products Administration for treating weight loss in individuals with obesity. Up to now, there is a paucity of research on the potential impact of GLP-1RAs on reproductive, maternal and perinatal outcomes in women with PCOS and obesity undergoing fertility treatment. Given its effectiveness as a weight loss medication, benalutide theoretically holds promise for enhancing reproductive outcomes in women with PCOS and obesity prior to fertility treatment by facilitating weight reduction.

ELIGIBILITY:
Inclusion Criteria:

Women with a wish to conceive; Women with PCOS (Rotterdam criteria); 28 kg/m2≤BMI<35kg/m2;

Exclusion Criteria:

Women with medical morbidity; Endocrine disorders; Abnormalities in liver and kidney function; Other medications such as glucocorticoids, anti-androgen drugs ;(spironolactone, cyproterone acetate, flutamide, etc.) within the last 3 months; Acute infections, severe cardiovascular disease, malignant tumors; Ongoing weight loss therapy (>5% weight loss in the last 3 months) or history of gastrointestinal surgery; Uterine anomalies or untreated tubal hydrosalpinx; Receiving a donor oocyte or donor sperm cycle; Chromosome abnormality or recurrent miscarriage; planning preimplantation genetic testing (PGT); Any other contraindications to fertility treatment; Allergic to or contraindicated for GLP-1 class medications.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 392 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 18 months

SECONDARY OUTCOMES:
BMI change from baseline to the 3rd month in kg/m2 | 3 months
Spontaneous resumption of ovulation | 3 months
Clinical pregnancy | 9 months
Ongoing pregnancy | 11 months
Pregnancy loss | 18 months
Gestational age at delivery | 18 months
Time to pregnancy leading to live birth | 18 months
Hypertensive disorders of pregnancy | 18 months
Gestational diabetes | 18 months
Birth weight in kg | 18 months
Neonatal mortality | 18 months
Major congenital anomaly | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided